CLINICAL TRIAL: NCT02432937
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Phase III Study of Corever for the Treatment of Hypertension
Brief Title: Corever in the Treatment of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSHCR1201
Record Dates: First submitted 2015-01-29; First posted 2015-05-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Corever; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Corever middle dose (Placebo Comparator)
  Interventions: Drug: Corever
- Corever high dose (Placebo Comparator)
  Interventions: Drug: Corever
- Placebo (Placebo Comparator)
  Interventions: Drug: Corever

INTERVENTIONS:
Drug: Corever — Corever
  Other Names: CRTA04

SUMMARY:
The study primarily aims to compare the effects of two doses of Corever with placebo in patients with hypertension.

DETAILED DESCRIPTION:
The study aims to compare the effects of two doses of Corever with placebo in patients with essential hypertension. Eligible subjects who belong to one of the following subtypes are planned to be enrolled: (1) patients with essential hypertension without drug control, or (2) uncontrolled hypertension despite treatment with up to 2 antihypertensive agents. Of note, the second category will receive randomized study treatments in addition to continuing their previous medication throughout the trial. The study also wants to investigate the safety profile of Corever during treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 20-90 years of age
2. Patients who belong to either one of the following categories:

   With essential hypertension, as measured by office BP and are not on antihypertensive treatment at screening .

   With uncontrolled hypertension despite treatment with up to 2 antihypertensive agents, and the type and dose of the agents shall be maintained for at least 28 days prior to entering this trial.
3. Agree to and are able to follow the study procedures.
4. Understand the nature of the study, and have signed informed consent forms.

Exclusion Criteria:

1. Patients with any of the following conditions:

   * Malignant hypertension
   * Secondary hypertension
   * Average sitting SBP ≥ 180 mmHg
   * Advanced hypertensive retinopathy
   * Type 1 diabetes
   * Acute coronary syndrome
   * Clinical significant valvular disease
   * Hypertrophic cardiomyopathies
   * New York Heart Association class III -IV congestive HF
   * Second or third degree atrioventricular block or history of sick sinus syndrome unless a pacemaker is in place
   * Atrial fibrillation
   * Sinus bradycardia (<60 bpm)
   * Asthma
   * Stroke within 3 months
   * Cancer with expected survival less than 3 years
   * A difference of > 20 mmHg for SBP or > 10 mmHg for DBP between arms at screening
   * Severe hepatic impairment
   * A history of a serious hypersensitivity reaction.
2. Patients with clinically significant abnormalities.
3. Patients with known contraindication to Corever.
4. Female patients who are pregnant or lactating.
5. 5. Male or female patients of child-bearing potential who do not agree to use an effective method of contraception during the study.
6. Patients is currently participating in any other clinical trial within 30 days
7. Patients need to be treated with the permitted medication.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Seated Office SBP reduction (SBP each visit-SBP visit 2) | 8 weeks
  To compare the change in office SBP measurements by cuff assessments after 8 weeks of treatment

SECONDARY OUTCOMES:
Seated Office DBP reduction (DBP each visit-DBP visit 2) | 8 weeks
  1. To compare the change in office DBP measurements by cuff assessments after 8 weeks of treatment
  2. To compare the percentage of subjects who achieve BP goal as measured by cuff assessments (140/90 mmHg) after 8 weeks of treatment

OTHER OUTCOMES:
Safety-Adverse events | 8 weeks
Safety-Changes in vital signs | 8 weeks
Safety-Changes in laboratory examinations | 8 weeks
Safety-Changes in electrocardiograms | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chern-En Chiang, M.D., Ph.D.,, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (8):
- Taiwan (8):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei